CLINICAL TRIAL: NCT02337465
Title: Integrated 3D X-ray and Ultrasound Guided Radiation Therapy of Soft Tissue Targets
Brief Title: KV-CBCT and Ultrasound Imaging in Guiding Radiation Therapy in Patients With Prostate, Liver, or Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE6Y14
Record Dates: First submitted 2015-01-09; First posted 2015-01-13 (Estimated); Results first posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Adult Liver Carcinoma; Malignant Pancreatic Neoplasm; Prostate Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Pancreatic Neoplasms; Prostatic Neoplasms | interventions — Cone-Beam Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Diagnostic (KV-CBCT, ultrasound-guided radiation therapy) (Experimental): Patients undergo 3-Dimensional Ultrasound-Guided Radiation Therapy prior to and during radiation therapy. Patients also undergo kilo-voltage Cone-Beam Computed Tomography prior to radiation therapy.
  Interventions: Device: Cone-Beam Computed Tomography; Radiation: 3-Dimensional Ultrasound-Guided Radiation Therapy

INTERVENTIONS:
Device: Cone-Beam Computed Tomography — Undergo kilo-voltage cone beam computed tomography
Radiation: 3-Dimensional Ultrasound-Guided Radiation Therapy — Undergo ultrasound-guided radiation therapy
  Other Names: 3D Ultrasound-Guided Radiation Therapy

SUMMARY:
This clinical trial studies if kilo-voltage cone beam computed tomography (KV-CBCT) and ultrasound imaging works in guiding radiation therapy in patients with prostate, liver, or pancreatic cancer. Computer systems, such as KV-CBCT and ultrasound imaging, allow doctors to create a 3-dimensional picture of the tumor may help in planning radiation therapy and may result in more tumor cells being killed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate the feasibility of combining on-board cone beam computed tomography (CBCT) with ultrasound imaging to overcome the shortcomings of CBCT or ultrasound imaging alone for imaging guided radiotherapy delivery.

OUTLINE:

Patients undergo ultrasound imaging prior to and during radiation therapy. Patients also undergo kilo-voltage cone beam computed tomography prior to radiation therapy.

Update (2021/02/04): Removed secondary outcome "Incidence of Adverse Events Related to the Ultrasound Probe". Per PI: Study initially intended to involve a non-FDA approved probe for use with liver patients but removed this section.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have either 1) cancer involving the liver by biopsy or radiographic criteria, or 2) prostate cancer by biopsy, with the intent of undergoing definitive dose radiation therapy to targets within the liver, or prostate. Patients with prostatectomy receiving post-operative radiotherapy are also eligible.
* Karnofsky performance status (PS) ≥ 70
* Subjects must have the ability to understand and the willingness to sign a written informational form

Exclusion Criteria:

* Patients with uncontrolled inter-current illness or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09-22 (Actual); Primary Completion 2019-12-14 (Actual); Study Completion 2019-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ping Xia, PhD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center; Kevin Stephans, MD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic (KV-CBCT, Ultrasound-guided Radiation Therapy)
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (KV-CBCT, Ultrasound-guided Radiation Therapy)
Number analyzed (Participants) | 30
Age, Customized [Count of Participants; unit: Participants]
  40-49 years | 1
  50-59 years | 2
  60-69 years | 12
  70-79 years | 14
  80-89 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Ultrasound Images Which Are Clinically Adequate for Treatment Set-up
Description: Percentage of ultrasound images which are clinically adequate for treatment set-up in the judgment of the treating physician
Time Frame: Up to 1 year
Population: Participants enrolled on study
Measure: Number; unit: Percent of images
Groups:
- Diagnostic (KV-CBCT, Ultrasound-guided Radiation Therapy): Participants undergo 3-Dimensional Ultrasound-Guided Radiation Therapy prior to and during radiation therapy. Participants also undergo kilo-voltage Cone-Beam Computed Tomography prior to radiation therapy.
  Cone-Beam Computed Tomography: Undergo kilo-voltage cone beam computed tomography
  3-Dimensional Ultrasound-Guided Radiation Therapy: Undergo ultrasound-guided radiation therapy
Arm/Group | Diagnostic (KV-CBCT, Ultrasound-guided Radiation Therapy)
Number analyzed (Participants) | 30
Percent of images | 100

2. Primary Outcome: Number of Participants Able to Have the Ultrasound Probe Attached During the Entire Treatment Course
Description: Proportion of participants able to have the ultrasound probe attached during the entire treatment course
Time Frame: Up to 1 year
Population: Participants enrolled on study
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic (KV-CBCT, Ultrasound-guided Radiation Therapy)
Number analyzed (Participants) | 30
Participants | 29

3. Primary Outcome: Percent of Patients Whose Plan Quality Was Not Not Affected in the Presence of the Ultrasound Probe
Description: Quality of plans for patients not affected in the presence of the ultrasound probe, defined as no more than a 2% decrease in tumor coverage, and also no more than a 2% increase in the dose to the most critical normal tissue for that tumor location
Time Frame: Up to 1 year
Population: Participants enrolled on study
Measure: Number; unit: percentage of participants
Arm/Group | Diagnostic (KV-CBCT, Ultrasound-guided Radiation Therapy)
Number analyzed (Participants) | 30
percentage of participants | 100

ADVERSE EVENTS:
Description: No plan to collect adverse event data (per-protocol)
Arm/Group | Diagnostic (KV-CBCT, Ultrasound-guided Radiation Therapy)
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT02337465/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT02337465/ICF_001.pdf